CLINICAL TRIAL: NCT05962125
Title: Effects of Three Open-lung Strategies on Respiratory Function and Lung Injury in Protective Ventilation for Laparoscopic Anterior Resection: a Randomized Controlled Trial
Brief Title: The Role of Periodic Alveolar Recruitment Maneuvers in Intraoperative Protective Ventilation
Acronym: REMAIN-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: E2023069
Record Dates: First submitted 2023-06-28; First posted 2023-07-27 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2023-09

CONDITIONS: Mechanical Power; Alveolar Recruitment Maneuvers; Protective Ventilation; Postoperative Pulmonary Complications
MeSH Terms: interventions — Positive-Pressure Respiration

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- periodic alveolar recruitment maneuvers (PARM) alone (Experimental): Alveolar recruitment maneuvers [ARM] repeated every 30 min after tracheal intubation and after any disconnection from the ventilator.
  Interventions: Other: periodic alveolar recruitment maneuvers
- positive end-expiratory pressure (PEEP) alone (Active Comparator): PEEP was routinely set at 6 cm H2O. If it was in a state of Trendelenburg position or carbon dioxide pneumoperitoneum, PEEP was set to 8 cm H2O.
  Interventions: Other: positive end-expiratory pressure
- a combination of PEEP and PARM (Active Comparator): Alveolar recruitment maneuvers [ARM] repeated every 30 min after tracheal intubation and after any disconnection from the ventilator. PEEP was routinely set at 6 cm H2O. If it was in a state of Trendelenburg position or carbon dioxide pneumoperitoneum, PEEP was set at 8 cm H2O.
  Interventions: Other: periodic alveolar recruitment maneuvers; Other: positive end-expiratory pressure

INTERVENTIONS:
Other: periodic alveolar recruitment maneuvers — A stepwise increment of tidal volume was used for each ARM.
  Arms: a combination of PEEP and PARM; periodic alveolar recruitment maneuvers (PARM) alone
Other: positive end-expiratory pressure — a PEEP of 6 to 8 cm H2O
  Arms: a combination of PEEP and PARM; positive end-expiratory pressure (PEEP) alone

SUMMARY:
The goal of this clinical trial is to compare three open-lung strategies on respiratory function and lung injury in protective ventilation for laparoscopic anterior resection. It aims to answer whether a periodic alveolar recruitment maneuvers (PARM) strategy alone was an appropriate open-lung strategy in intraoperative protective ventilation. Patients were randomly assigned (1:1:1) to receive one of three open-lung strategies in protective ventilation: PARM alone (alveolar recruitment maneuvers [ARM] repeated every 30 min), positive end-expiratory pressure (PEEP) alone (a PEEP of 6 to 8 cm H2O), or a combination of PEEP and PARM (a PEEP of 6 to 8 cm H2O combined with ARM repeated every 30 min). The primary outcome is the mechanical power before the end of intraoperative mechanical ventilation. Secondary outcomes included the accumulative intraoperative mechanical power, an arterial partial pressure of oxygen (PaO2) / inhaled oxygen concentration (FiO2) ratio (P/F ratio) before the end of intraoperative mechanical ventilation, the rates of respiratory failure at post-anesthesia care unit (PACU) and three postoperative days, the concentration of soluble advanced glycation end products receptor (sRAGE) and Clara cell protein 16 (CC16) at the end of surgery, postoperative pulmonary complications score, postoperative hospitalization days and so on.

ELIGIBILITY:
Inclusion Criteria:

1. Undergoing elective laparoscopic anterior resection and expected duration of mechanical ventilation 2 to 5 h.
2. Had an intermediate risk of developing postoperative pulmonary complications.
3. Pulse oxygen saturation in room air ≥ 94%.
4. Aged 60 to 80 years.

Exclusion Criteria:

* 1. Had received invasive mechanical ventilation for longer than 1 h within the last 2 weeks prior to surgery.

  2. Had a history of pneumonia within 1 month prior to surgery. 3. Had severe chronic obstructive pulmonary disease or pulmonary bullae. 4. Had a progressive neuromuscular illness. 5. With an American Society of Anesthesiologists (ASA) physical status of IV or higher.

  6. Intracranial hypertension. 7. Body mass index (BMI) ≥30 kg/m2. 8. Were involved in other interventional studies.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2023-08-21 (Actual); Primary Completion 2023-11-08 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Intraoperative mechanical power | Before the end of intraoperative mechanical ventilation, about 5 to 10 minutes before the end of surgery
  Intraoperative mechanical power, calculated from values of tidal volume (Vt ), respiratory rate (RR), positive end-expiratory pressure (PEEP), plateau pressure (Pplat), and peak inspiratory pressure (Ppeak), using the following formula: mechanical power (J/min) = 0.098 × RR × Vt × (PEEP + ½[Pplat - PEEP] + [Ppeak - Pplat])

SECONDARY OUTCOMES:
Mechanical power during capnoperitoneum | 30 minutes after starting carbon dioxide pneumoperitoneum
  mechanical power, J/min
Accumulative mechanical power (AMP) | During intraoperative mechanical ventilation, an average of 3 hours
  Accumulative mechanical power (AMP) = AMP before capnoperitoneum + AMP during capnoperitoneum + AMP after capnoperitoneum. Accumulative mechanical power before capnoperitoneum = mechanical power before capnoperitoneum (10 min after mechanical ventilation) × the length of mechanical ventilation before capnoperitoneum. Accumulative mechanical power during capnoperitoneum = mechanical power during capnoperitoneum (30 min after mechanical ventilation) × the length of mechanical ventilation during capnoperitoneum. Accumulative mechanical power after capnoperitoneum (after the end of capnoperitoneum) = mechanical power after capnoperitoneum (10 min after the end of capnoperitoneum) × the length of mechanical ventilation after capnoperitoneum
An arterial partial pressure of oxygen (PaO2) / Inhaled oxygen concentration (FIO2) ratio (P/F ratio) | Before the end of intraoperative mechanical ventilation, about 5 to 10 minutes before the end of surgery
  P/F ratio, mmHg
Shunt fraction | Before the end of intraoperative mechanical ventilation, about 5 to 10 minutes before the end of surgery
  Shunt fraction, %
Dead space rate | Before the end of intraoperative mechanical ventilation, about 5 to 10 minutes before the end of surgery
  Arterial carbon dioxide partial pressure (PaCO2); partial pressure of carbon dioxide in end expiratory gas (PetCO2); Dead space fraction = (PaCO2-PetCO2)/ PaCO2.
Rate of respiratory failure at post-anesthesia care unit (PACU) | Stay in the PACU for at least 20 minutes and at most 3 hours; assessed at 5 to 10 minutes before leaving PACU
  Respiratory failure: PaO2 < 60 mmHg or pulse oxygen saturation (SpO2) < 90% on room air, or a P/F ratio < 300 mmHg and requiring oxygen therapy.
Soluble advanced glycation end products receptor (sRAGE) | 20 minutes after entering PACU
  The concentration of plasma sRAGE, pg/ml
Clara cell protein 16 (CC16) | 20 minutes after entering PACU
  The concentration of plasma CC16, ng/ml
Surfactant Protein D (SP-D) | 20 minutes after entering PACU
  The concentration of plasma SP-D, ug/ml
Interleukin 6 (IL-6) | 20 minutes after entering PACU
  The concentration of plasma IL-6, pg/ml
Rate of postoperative respiratory failure | Time Frame: Day 0 to 3 after surgery
  Respiratory failure: PaO2 < 60 mmHg or SpO2 < 90% on room air, or a P/F ratio < 300 mmHg and requiring oxygen therapy.
Rate of sustained hypoxaemia | Day 0 to 3 after surgery
  Sustained hypoxaemia, hypoxaemia at any two consecutive days; hypoxaemia: during a follow-up visit when the patient was awake and breathing room air, SpO2 ≤ 92% or the change of SpO2 (ΔSpO2, preoperative SpO2 minus postoperative SpO2) ≥ 5%.
Postoperative pulmonary complications score | Day 0 to 3 after surgery
  Postoperative pulmonary complications score: Operational Definitions of Postoperative Pulmonary Complications (Doi: 10.1001/jama.296.15.1851), graded on a scale from 0 (no pulmonary complications) to 4 (the most severe complications).
Postoperative hospitalization days | Day 0 to 30 after surgery
  The duration between the operation date and the actual discharge date.
Death from any cause | Day 0 to 30 after surgery
  Intraoperative or postoperative death from any cause
Rate of intraoperative hypotension | During intraoperative mechanical ventilation, an average of 3 hours
  Intraoperative hypotension, mean arterial pressure (MAP) < 60 mmHg lasting more than 3 minutes.
Rate of need for vasoconstrictors | During intraoperative mechanical ventilation, an average of 3 hours
  MAP < 60 mmHg and using any vasoconstrictors.
Rate of intraoperative hypoxemia | During intraoperative mechanical ventilation, an average of 3 hours
  Intraoperative hypoxemia, SpO2 ≤ 92% lasting more than 3 minutes.
Rate of intraoperative bradycardia | During intraoperative mechanical ventilation, an average of 3 hours
  Intraoperative bradycardia, heart rate ≤ 50 bpm and the decrease of heart rate from the basic value ≥ 20% lasting more than 3 minutes.
Rate of pneumothorax | During surgery or within 7 days after surgery
  Pneumothorax, air in the pleural space with no vascular bed surrounding the visceral pleura.
Rate of pleural effusion | within 7 days after surgery
  Pleural effusion, diagnosed according to previous literature (Doi: 10.1097/EJA.0000000000000118).
Unexpected admission to ICU | within 30 days after surgery
  It does not include the patients who enter ICU at the request of surgeons but have normal spontaneous breathing, stable circulation and no disturbance of consciousness.
Tumor Necrosis Factor alpha (TNF-α) | 20 minutes after entering PACU
  TNF-α, pg/ml.

CONTACTS AND LOCATIONS:
Overall Officials: Hong Li, MD, Principal Investigator — The Sixth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- The Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China